CLINICAL TRIAL: NCT05166512
Title: Development and Pilot Evaluation of a Novel Cooking Skills Intervention to Prevent Diabetes
Brief Title: Pilot Trial of a Novel Cooking Skills Intervention (DPPCooks) to Prevent Diabetes
Acronym: DPPCooks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00018839; K01DK119166 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard DPP (Active Comparator): Standard DPP (over 12 months)
  Interventions: Behavioral: DPP
- DPP Cooks (Experimental): Standard DPP plus DPP Cooks (over 12 months, with 6 active cooking sessions during the first 4 months)
  Interventions: Behavioral: DPP Cooks

INTERVENTIONS:
Behavioral: DPP Cooks — 6 'food agency' based cooking skills classes during the first 4 months of the DPP
  Arms: DPP Cooks
Behavioral: DPP — Standard DPP
  Arms: Standard DPP

SUMMARY:
In this pilot trial participants will be randomized 1:1 to participate in either standard Diabetes Prevention Program (DPP) vs. DPP plus a novel cooking skills intervention (DPP Cooks). The researchers hypothesize that participants randomized to DPP Cooks will have greater weight loss, better diet quality at 4 months, and greater confidence in their cooking skills and ability to implement dietary changes recommended in the DPP.

DETAILED DESCRIPTION:
This study is a randomized pilot trial testing a novel cooking skills intervention (DPP Cooks) vs. the standard Diabetes Prevention Program (DPP). The DPP is a widely disseminated evidenced-based lifestyle behavior change program to help adults with pre-diabetes lose weight and prevent type-2 diabetes. In this trial the investigators will test whether the addition of food-agency based cooking skills classes improves the effectiveness of the DPP. This trial will take place in Baltimore, MD in collaboration with community partner DPP providers. The trial has been informed by formative work with prior DPP participants and has used a Community Based Participatory Research (CBPR) approach to developing the DPP Cooks intervention. Participants will be randomized 1:1 to participate in either standard DPP vs. DPP Cooks. The length of the trial will be 12 months and outcomes will be measured at baseline, 4 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults in Baltimore City
* eligible for DPP based on Centers for Disease Control guidelines
* possession of a smart phone with camera
* can commit to 12 month study participation

Exclusion Criteria:

* current or prior diagnosis of type 1- or type 2 diabetes
* non-English speaker
* participating in another research study that may effect diabetes, diet, or weight loss
* currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Wolfson, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Brancati Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Randomized
Arm/Group | Standard DPP | DPP Cooks
Started | 22 | 23
Completed | 19 | 23
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Baseline Data Collection
Arm/Group | Standard DPP | DPP Cooks
Started | 19 | 23
DPP Session 0 | 19 | 23
DPP Session 1 | 18 | 20
Completed | 16 | 20
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0
Period: 4 Month Data Collection
Arm/Group | Standard DPP | DPP Cooks
Started | 16 | 20
Completed | 14 | 15
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Period: 12 Month Data Collection
Arm/Group | Standard DPP | DPP Cooks
Started | 14 | 15
Completed | 10 | 14
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: participants who had baseline data collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard DPP | DPP Cooks | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.8) | 56.5 (17.2) | 55.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 20 | 36
Education [Count of Participants; unit: Participants]
  some high school | 1 | 0 | 1
  high school | 6 | 2 | 8
  some college | 3 | 6 | 9
  college graduate | 6 | 12 | 18
Marital Status [Count of Participants; unit: Participants]
  single | 6 | 4 | 10
  married | 3 | 7 | 10
  living with partner | 1 | 3 | 4
  divorced, separated, widowed | 6 | 6 | 12
Income [Count of Participants; unit: Participants]
  <$35,000/ year | 6 | 7 | 13
  #35,000-$59,000/ year | 6 | 5 | 11
  $60,000-$85,000/ year | 1 | 5 | 6
  >$85,000/ year | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Absolute Body Weight (Kilograms (kg))
Description: Weight change will be measured in absolute kg. Weight will be measured at baseline, 4 months and 12 months. Weight will be measured by DPP coaches at weekly meetings (or, if DPP groups are meeting virtually, weight will be reported by participants to their DPP coaches in weekly virtual meetings).
Time Frame: baseline, 4 months and 12 months
Population: Change from baseline to 4 months includes the 29 individuals who completed 4 month data collection. Change from baseline to 12 months includes the 24 individuals who completed 12 month data collection.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
kg
  change from baseline to 4 months | -2.12 (1.61) | -1.00 (1.55)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | -5.27 (1.67) | -4.15 (1.57)

2. Primary Outcome: Change From Baseline in Percentage of Baseline Bodyweight
Description: Weight change will be measured in the percent of body weight change. Weight will be measured at baseline, 4 months and 12 months. Weight will be measured by DPP coaches at weekly meetings (or, if DPP groups are meeting virtually, weight will be reported by participants to their DPP coaches in weekly virtual meetings).
Time Frame: baseline, 4 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of body weight
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
percentage of body weight
  change from baseline to 4 months | -1.96 (1.49) | -0.95 (1.44)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | -5.12 (1.55) | -4.11 (1.46)

3. Secondary Outcome: Difference From Baseline in Diet Quality (Healthy Eating Index- 2015) Score
Description: Dietary intake and diet quality (Healthy Eating Index (HEI-2015) as measured by the Remote Food Photography Method (RFPM) over 3 days of dietary intake at baseline and 4 months. The HEI-2015 is a score from 0-100 with high score indicating better diet quality. The HEI-2015 measures how well an individuals dietary intake aligns with the 2015 US Dietary Guidelines.
Time Frame: Baseline and at 4 months
Population: all individuals with data at baseline and 4 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
score on a scale | 1.52 (3.50) | -2.81 (3.37)

4. Secondary Outcome: Change From Baseline in Cooking Confidence
Description: Cooking confidence, attitudes and behaviors will be measured via online survey (7- point Likert Scale (strongly agree to strongly disagree) questions) at baseline, 4 months and 12 months. Survey items were based on prior literature, but there is not a formal named scale that was used. Cooking confidence was assessed by 7 items all measured on a 7 point Likert scale. Negative items were reverse coded, then 7 confidence items were summed to create a overall confidence score (range 7-49) with higher values indicating higher confidence.
Time Frame: baseline, 4 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
units on a scale
  change from baseline to 4 months | 0.84 (1.37) | 0.47 (1.31)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | 1.84 (1.44) | 1.46 (1.33)

5. Secondary Outcome: Change From Baseline in Food Agency Measured Via the Cooking and Food Provisioning Action Scale (CAFPAS)
Description: The Cooking and Food Provisioning Action Scale (CAFPAS) is a 28 question scale in which higher scores indicate higher Food Agency. All questions in the CAFPAS are measured on 7-point Likert Scales (strongly agree to strongly disagree). The CAFPAS has 3 sub-scales which are scored by summing the scores on each individual question (after reverse coding negative items) and are then standardized. Then the 3 standardized sub-scale scores are summed to generate an overall CAFPAS score in which higher scores indicate better Food Agency. In this sample scores range from 10.48- 22.25 points with higher scores indicating better Food Agency.
Time Frame: baseline, 4 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: change in score on a scale
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
change in score on a scale
  change from baseline to 4 months | 0.16 (0.42) | -0.53 (0.41)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | 0.93 (0.44) | 0.24 (0.41)

6. Secondary Outcome: Participant Food Security Status Over the Past 30 Days Using the 10-item United States Department of Agriculture (USDA) Adult Food Security Survey Module
Description: The USDA Adult Food Security Survey Module is a 10-item progressive survey instrument in which individuals are asked about the food situation in their household over the last 30 days. Scores are summed and generate the following categories: High food security status (raw score: 0), Marginal food security status (raw score: 1-2), Low food security status (raw score 3-5), Very low food security status (raw score: 6-10).
Time Frame: baseline, 4 months and 12 months
Population: Analyzed among all participants enrolled and at each time point. One participant still enrolled at 12 months was missing data for food insecurity.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 16 | 20
Participants
  Baseline: High food security | 9 | 11
  Baseline: Marginal food security | 5 | 4
  Baseline: Low food security | 1 | 5
  Baseline: Very low food security | 1 | 0
  4 months: number analyzed (Participants) | 14 | 15
  4 months: High food security | 10 | 6
  4 months: Marginal food security | 3 | 2
  4 months: Low food security | 1 | 3
  4 months: Very low food security | 0 | 4
  12 months: number analyzed (Participants) | 10 | 13
  12 months: High food security | 8 | 5
  12 months: Marginal food security | 2 | 3
  12 months: Low food security | 0 | 2
  12 months: Very low food security | 0 | 3

7. Secondary Outcome: Change From Baseline in Cooking Attitudes
Description: Cooking confidence, attitudes and behaviors will be measured via online survey (7- point Likert Scale (strongly agree to strongly disagree) questions) at baseline, 4 months and 12 months. Survey items were based on prior literature, but there is not a formal named scale that was used. Attitudes were assessed by 11 questions all scored on a 7 point Likert scale. Negative attitudes were reverse coded, then scores were summed across all 11 items to create an overall Attitudes score (range: 7-77) with higher scores indicating more positive attitudes about cooking.
Time Frame: baseline, 4 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
units on a scale
  change from baseline to 4 months | 1.57 (1.85) | -0.28 (1.76)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | 3.92 (1.89) | 2.07 (1.77)

8. Secondary Outcome: Change From Baseline in Cooking Behavior (Days Cooking Dinner)
Description: Cooking confidence, attitudes and behaviors will be measured via online survey (7- point Likert Scale (strongly agree to strongly disagree) questions) at baseline, 4 months and 12 months. To assess behavior change, an item from the National Health an Nutrition Examination Survey (NHANES) assessing frequency of cooking dinner was used. Change in number of days (0-7) cooking is reported with higher numbers indicating more frequent cooking dinner at home.
Time Frame: baseline, 4 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard DPP | DPP Cooks
Number analyzed (Participants) | 14 | 15
days
  change from baseline to 4 months | 0.80 (0.39) | 0.43 (0.38)
  change from baseline to 12 months: number analyzed (Participants) | 10 | 14
  change from baseline to 12 months | 0.86 (0.41) | 0.49 (0.38)

9. Other Pre Specified Outcome: Program Attendance Among DPP and DPP Cooks Participants
Description: DPP coaches will report weekly session attendance for all trial participants. Attendance at a higher number of sessions will be a favorable result.
Time Frame: 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Program Satisfaction Among DPP Cooks Participants (Qualitative)
Description: Investigators will use interviews or focus groups with DPP Cooks participants to gather qualitative feedback about program satisfaction among participants
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Standard DPP | DPP Cooks
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT05166512/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05166512/ICF_000.pdf